CLINICAL TRIAL: NCT01579994
Title: A Phase I Study of Crizotinib and Ganetespib (STA-9090) in ALK Positive Lung Cancers
Brief Title: Crizotinib and Ganetespib (STA-9090) in ALK Positive Lung Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-015
Record Dates: First submitted 2012-04-16; First posted 2012-04-18 (Estimated); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Advanced Lung Cancer
Keywords: adenocarcinoma; Lung; Metastatic; Crizotinib; Ganetespib; STA-9090; ALK Positive Lung Cancers; 12-015
MeSH Terms: conditions — Adenocarcinoma; Neoplasm Metastasis | interventions — STA 9090; Crizotinib

ARMS (1):
- Ganetespib (STA-9090) and crizotinib (Experimental): This protocol is a phase I single arm, open label, single institution study of crizotinib and ganetespib (STA-9090) in patients with ALK+ advanced NSCLC who are crizotinib naïve.
  Interventions: Drug: Ganetespib (STA-9090) and crizotinib

INTERVENTIONS:
Drug: Ganetespib (STA-9090) and crizotinib — Ganetespib (STA-9090) is given intravenously (days 1 and 8 of a 21 day cycle). Crizotinib will be given at the FDA approved dose of 250mg orally twice daily in a continuous fashion.

SUMMARY:
About 18 patients will take part in the phase 1 portion of the trial. In the beginning of the study, 3 patients will be treated with a low dose of ganetespib (STA-9090) and the standard dose of crizotinib. If this dose does not cause significant side effects, it will be increased as new patients take part in the study. The study will only be open at Memorial Sloan Kettering Cancer Center.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven diagnosis confirmed at MSKCC of advanced lung adenocarcinoma that is locally advanced or metastatic (stage III/IV).
* Positive for translocation or inversion events involving the ALK gene locus as determined standard methods (including but not limited to by FISH and IHC testing).
* No prior treatment with crizotinib, but they may have received prior cytotoxic chemotherapy.
* Age ≥ 18 years.
* Measurable (RECIST 1.1) indicator lesion not previously irradiated.
* Karnofsky Performance Status ≥ 70%
* Able to take oral medications
* A negative serum pregnancy test obtained within two weeks prior to administration of the experimental agents in all pre-menopausal women (last menstrual period ≤ 24 months ago).
* All women of child bearing potential (WOCBP) and sexually active men must agree to use adequate methods of birth control throughout the study which include use of oral contraceptives with an additional barrier method, double barrier methods (diaphragm with spermicidal gel or condoms with contraceptive foam), Depo-Provera, partner vasectomy and/or tubal libation and total abstinence.

Exclusion Criteria:

* Prior crizotinib therapy
* Inadequate recovery from any toxicity related to prior treatment (to Grade 1 or baseline).
* Inadequate hematologic function defined as:

  * Absolute neutrophil count (ANC) < 1,000 cells/mm³.
  * Platelet count < 75,000/mm³
  * Hemoglobin < 9.0g/dL.

Inadequate hepatic function defined by:

* AST and/or ALT > 3x upper limited of normal (ULN).
* Total bilirubin > 2x ULN.
* Alkaline phosphatase > 3x ULN.
* Patients with hepatic metastases may have ALT/AST ≤ 5x ULN.
* Patients with hepatic and/or bone metastases may have an AP ≤ 5x ULN.
* Inadequate renal function defined by serum creatinine > 2x ULN Uncontrolled systemic fungal, bacterial, viral or other infection (defined as exhibiting ongoing signs/symptoms related to infection without improvement, despite appropriate anti-infective medications or other treatment).
* Patients with clinically active brain metastasis (requiring therapy with steroids or radiation therapy). Patients with clinically stable brain metastases (previously treated or untreated) for two weeks are eligible.
* Significant cardiac disease (e.g. New York Heart Association (NYHA) Class 3 or 4; myocardial infarction within the past 6 months; unstable angina; coronary angioplasty or coronary artery bypass graft (CABG) within the past 6 months; or uncontrolled atrial or ventricular cardiac arrhythmias).
* Previously or current malignancies at other sites within the last 2 years, with the exception of adequately treated in situ carcinoma of the cervix, basal or squamous cell carcinoma of the skin, or prostate cancer that does not require active treatment per National Comprehensive Cancer Network (NCCN) guidelines.
* Women who are pregnant or lactating
* Use of drugs or food that are known potent CYP3A4 inhibitors (see Appendix C)
* Use of drugs that are known potent CYP3A4 inducers (see Appendix D)
* Any other condition that, in the opinion of the Investigator, may compromise the safety, compliance of the patient, or would preclude the patient from successful completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2012-04-16 (Actual); Primary Completion 2020-12-28 (Actual); Study Completion 2020-12-28 (Actual)

PRIMARY OUTCOMES:
maximum tolerated dose | 1 year
  A standard 3+3 design will be used to find the maximum tolerated dose (MTD). Patients who withdraw before completing a full cycle will be replaced. There will be three set dose levels, using the approved dose of crizotinib, with 50%, 75% and 100% of the ganetespib (STA-9090) maximum tolerated dose of 200 mg/m2.
efficacy | 1 year
  patients with ALK rearranged NSCLC at delaying acquired resistance to crizotinib by measuring progression free survival

SECONDARY OUTCOMES:
overall survival (OS) | 1 year
  as defined by time from study entry to death due to any cause and overall response rate (RR), as defined by the combination of complete responses and partial responses according to RECIST 1.1
safety profile | 2 years
  Toxicity will be graded according to the NCI Common Terminology Criteria for Adverse Events (NCI CTCAE), version 4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Gregrory Riely, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - Memoral Sloan Kettering Cancer Center, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering at Mercy Medical Center, Rockville Centre, New York
  - Memoral Sloan Kettering Cancer Center at Phelps, Sleepy Hollow, New York

REFERENCES:
- [Derived] Wong KM, Noonan S, O'Bryant C, Jimeno A. Alectinib for the treatment of ALK-positive stage IV non-small cell lung cancer. Drugs Today (Barc). 2015 Mar;51(3):161-70. doi: 10.1358/dot.2015.51.3.2294597. PMID 25876560
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/